CLINICAL TRIAL: NCT05225428
Title: Video Education With Result Dependent dIsclosure
Acronym: VERDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Huma Rana, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-508; R01HG011928 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-02-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Genetic Testing; Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Colorectal Cancer; Renal Cancer; Melanoma; Sarcoma
Keywords: Genetic Testing; Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Colorectal Cancer; Renal Cancer; Melanoma; Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Kidney Neoplasms; Melanoma; Sarcoma | interventions — Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QUALITATIVE ASSESSMENT (Experimental): This part of the research study involves watching a brief educational video about genetic testing for inherited cancer risk (about 8 minutes) before completing a short interview by video or telephone with trained researchers. This interview will be digitally recorded for later review.
  It is expected that about 20 people will take part in this part of the research study.
  In the larger part of the study that will happen after this part of the study, it is expected 1000 people will participate.
  Interventions: Behavioral: Video Education
- RCT-VERDI (Experimental): A randomized controlled trial (RCT) will evaluate the VERDI model vs. standard genetic counseling
  Interventions: Behavioral: Video Education
- RCT-Genetic Counseling (Experimental): A randomized controlled trial (RCT) will evaluate the VERDI model vs. standard genetic counseling
  Interventions: Behavioral: Genetic Counseling

INTERVENTIONS:
Behavioral: Video Education — Investigator-developed, professionally animated and produced 8-minute video (Video Education) summarizing the core educational components of a genetic counseling visit
  Other Names: VERDI
  Arms: QUALITATIVE ASSESSMENT; RCT-VERDI
Behavioral: Genetic Counseling — Standard genetic counseling
  Arms: RCT-Genetic Counseling

SUMMARY:
The overall study objective of this trial study is to identify and evaluate strategies to improve the accessibility of the video education with result dependent disclosure (VERDI) model, increasingly utilized as a pre-genetic testing (pretest) education alternative in clinical practice, to better serve a more diverse patient population at risk for hereditary cancers.

DETAILED DESCRIPTION:
This study consists of two parts:

* Qualitative assessment:

  * This part of the research study involves watching a brief educational video about genetic testing for inherited cancer risk (about 8 minutes) before completing a short interview by video or telephone with trained researchers. This interview will be digitally recorded for later review. Participation in the study will be considered complete after the interview is finished. The qualitative assessment study will recruit 20 total participants.
  * The data gathered from this study will inform the refinement and adaptation of the VERDI model for the subsequent randomized controlled trial.
* Randomized control trial:

  * A randomized controlled trial (RCT) will evaluate the VERDI model vs. standard genetic counseling in 1000 participants

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Current or prior diagnosis of breast cancer, ovarian cancer, pancreatic cancer, prostate cancer, colorectal cancer, renal cancer, melanoma, or sarcoma
* Ability to understand spoken or written English or Spanish in a healthcare context
* Ability to understand and the willingness to sign a written informed consent document
* Black or Latinx (qualitative assessment study only)

Exclusion Criteria:

* Prior cancer genetic testing
* Prior germline genetic testing
* Active hematologic malignancy (e.g. chronic lymphocytic leukemia)
* Currently pregnant
* Currently incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Video Education Acceptability (Qualitative Interview Study) | 3 Weeks
  Pre- and post-test of knowledge of hereditary cancer risk and cancer genetic counseling with qualitative patient interview question domains and instruments to assess understanding of language and imagery of video education as correlated with measures of health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Q. Rana, MD., MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu